CLINICAL TRIAL: NCT02764567
Title: Essential Oil Aromatherapy Intervention: Easing the Discomforts of Phlebotomy With Essential Oil Aromatherapy
Brief Title: Essential Oil Aromatherapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthEast Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE 16 04 002
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Phobia Phlebotomy
MeSH Terms: interventions — Oils, Volatile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aromatherapy (Experimental): The participants randomized to aromatherapy will be offered one of three essential oils, 'applied' to their smell zone via cotton ball that are known to have anti-anxiety effect. These are:
  * ginger
  * calming
  * lavender The participant's choice will be documented in a database. The participant can chose an oil each time (i.e., they are not bound to use only the first choice oil). Pain and anxiety will be measured prior to receiving the essential oils and again after the phlebotomy procedure. Blood pressure and pulse will also be measured post-phlebotomy.
  Interventions: Other: Essential Oil
- Standard of Care (No Intervention): The participants randomized to standard of care will proceed to the outpatient phlebotomy room in the Heart Care Clinic as per usual care. Pain, anxiety, blood pressure and pulse will be assessed pre and post-procedure.

INTERVENTIONS:
Other: Essential Oil — Participants in this arm will be offered one of three essential oils: ginger, lavender or calming
  Arms: Aromatherapy

SUMMARY:
Lab sampling for clinical trial participants can be a stressful and painful experience. Most trial participants will have blood drawn for lab samples at multiple study visits. The participants must fast for up to ten hours before the blood sampling, in many cases, and patients often report a painful experience if more than one venipuncture occurs. In addition, the number of collection tubes can increase the anxiety level of the patient and the phlebotomist.

This project proposes to evaluate if essential oil aromatherapy results in less pain and /or anxiety when compared to usual care.

DETAILED DESCRIPTION:
The process of drawing blood for can be painful and stressful for any patient. Those patients who participate in a clinical trial agree to frequent lab sampling to monitor for effect and safety of the investigational product. The frequency is variable, from several times a day for a participant in the hospital to annually for some trials. Participants have reported anxiety regarding the number of tubes to be drawn, even resulting in near syncope, and pain with the venipuncture process.

The clinical trial nurses at HealthEast have utilized a variety of therapeutic techniques to ease the pain and anxiety experienced by the trial subjects, such as redirection, deep breathing, hand massage and guided imagery. These techniques have not been evaluated for effectiveness in easing pain and anxiety nor have they been compared with no intervention to determine if any intervention was more efficacious in alleviating pain and/or anxiety.

The primary objective of this study is determine if aromatherapy with an essential oil has a higher reported effect in anxiety and pain relief with venipunctures than standard of care (no therapy) among participants in HealthEast Clinical Trials Office studies.

Secondary objectives include comparing the number of venipunctures and blood collection tubes in the treatment arms.

This is a randomized, open label, prospective single site study designed to determine the effect of essential oil aromatherapy compared to usual care on pain and anxiety associated with venipunctures for clinical trial participants in the HealthEast Heart Care Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age
2. Must be currently participating in a clinical trial at HealthEast

Exclusion Criteria:

1. Known allergy to any of the oils used for aromatherapy
2. Less than age 18
3. Declined to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain Scores | At the time of study enrollment and again upon completion at 6 months
Change in Anxiety Scores | At the time of study enrollment and again upon completion at 6 months

SECONDARY OUTCOMES:
Number of venipunctures needed to collect required sample | At the time of study completion at 6 months
Number of blood collection tubes required for sample | At the time of study completion at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth Jorgeonson, RN, BSN, Principal Investigator — HealthEast Care System
Locations (1):
- HealthEast Clinical Trials Office, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be shared with the organization and submitted for publication. Individual participant data will not be shared.

REFERENCES:
- See also: Healing scents. (2015). Retrieved 12/23, 2015 — http://healingscents.net/blogs/learn/18685859-history-of-essential-oils
- See also: Tissearnd, R. (2011). Gattefossé's burn. Retrieved 12/23, 2015 — http://roberttisserand.com/2011/04/gattefosses-burn/